CLINICAL TRIAL: NCT03950271
Title: Phase II Clinical Study of PD1 Antibody (SHR-1210) Combined With Trastuzumab, Oxaliplatin and Capecitabine for Neoadjuvant Therapy of Gastric Adenocarcinoma/Gastroesophageal Junction Adenocarcinoma
Brief Title: SHR-1210 Combined With Trastuzumab , Oxaliplatin and Capecitabine for Neoadjuvant Therapy of Gastric Adenocarcinoma/Gastroesophageal Junction Adenocarcinoma
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Henan Cancer Hospital (Other Government)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: GCCG7
Record Dates: First submitted 2019-05-13; First posted 2019-05-15 (Actual); Last update posted 2024-02-28 (Actual); Status verified 2024-01

CONDITIONS: Gastric Cancer
MeSH Terms: conditions — Stomach Neoplasms | interventions — Trastuzumab; Oxaliplatin; Capecitabine

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- SHR-1210+ Trastuzumab + Oxaliplatin + Capecitabine (Experimental): trastuzumab + SHR-1210 + capecitabine + oxaliplatin for neoadjuvant chemotherapy 4-cycle.Then D2 radical surgery. The patients continued to receive capecitabine plus oxaliplatin for adjuvant therapy, and the total number of chemotherapy cycles was 8 cycles.
  Interventions: Drug: SHR-1210 Combined With Trastuzumab , Oxaliplatin and Capecitabine

INTERVENTIONS:
Drug: SHR-1210 Combined With Trastuzumab , Oxaliplatin and Capecitabine — 1. Neoadjuvant chemotherapy： SHR-1210 (200mg, d1, q3w) + trastuzumab ( 8 mg/kg on day 1 of the first cycle, followed by 6 mg/kg every 3 weeks) + capecitabine (1000mg/m2 bid d2-15, q3w) + Oxaliplatin (130mg/m2, d2, q3w)；4cycle
  2. postoperative adjuvant chemotherapy： Capecitabine (1000mg/m2 bid d1-14, q3w) + oxaliplatin (130mg/m2, d1, q3w)；The total number of chemotherapy cycles is 8 cycles.

SUMMARY:
The aim of this study is to observe the efficacy and safety of immume checkpoint inhibitor PD-1 SHR1210 combined with Trastuzumab , Oxaliplatin and Capecitabine for Neoadjuvant Therapy of locally advanced resectable gastric and gastroesophageal junction adenocarcinoma.

DETAILED DESCRIPTION:
This study is a prospective, one-arm, phase II clinical study to evaluate the safety and efficacy of SHR-1210 in combination with trastuzumab plus oxaliplatin and capecitabine for HER2-positive locally advanced resectable gastric adenocarcinoma and gastroesophageal junction adenocarcinoma during the perioperative treatment.

ELIGIBILITY:
Inclusion Criteria:

1. Signed the informed consent form
2. 18-75 years old
3. Pathologically confirmed gastric adenocarcinoma or gastroesophageal junction adenocarcinoma (cT4 or / and N+M0, MDT believes that perioperative treatment is required):

   1. No peritoneal metastasis in CT
   2. evaluated as a resectable lesion. Note: Whether there is a distant metastasis should be confirmed by CT or MR scan. If bone metastasis is suspected, a bone scan should be performed. If there is suspected peritoneal metastasis, a laparoscopy should be performed. If brain metastasis is suspected, CT or MR examination should be performed.
4. Have not received cytotoxic chemotherapy or targeted therapy and local tumor resection
5. HER2 immunohistochemistry 3+ and fluorescence in situ hybridization showed significant amplification
6. ECOG≤1
7. Tumor specimens that can be used to detect PD-L1 and MSI status can be provided. Detection of PD-L1 and MSI will be performed after enrollment. This test requires patients to provide paraffin-embedded biopsy specimens.
8. White blood cells ≥ 4×109/L, platelets without blood transfusion ≥ 100×109/L, absolute neutrophil count (ANC) ≥ 1.5×109/L without granulocyte stimulating factor, hemoglobin ≥ 90 g/L
9. bilirubin ≤ 1.5 times the upper limit of normal value, cereal grass and alanine aminotransferase ≤ 2.5ULN. If there is liver metastasis, the grass and alanine aminotransferase ≤ 5ULN.
10. serum creatinine ≤ 1.5ULN, or GFR > 45 ml / min
11. serum albumin ≥ 25 g / L (2.5 g / dL)
12. INR or APTT ≤ 1.5 ULN
13. Hepatitis B surface antigen positive patients need to detect hepatitis B DNA virus quantitative detection, only patients below the upper limit of normal detection can be enrolled, and long-term use ofanti-hepatitis B virus drugs

Exclusion Criteria:

1. Allergic to any test drug and its excipients, or have a history of severe allergies, or a contraindication to test drugs
2. Have a history of autoimmune disease or be active
3. Previously received allogeneic bone marrow transplantation or organ transplantation
4. Congenital pulmonary fibrosis, drug-induced pneumonia, organizing pneumonia, or CT-confirmed active pneumonia
5. HIV test positive
6. Active hepatitis B or hepatitis C
7. Active tuberculosis
8. Uncontrolled cancer pain
9. A live attenuated vaccine is injected within 4 weeks before the start of the study, or it is expected that a live attenuated vaccine will be injected within 5 months after the trial or the end of the trial.
10. Previous use of immunotherapy, including CTLA4, anti-PD-1, or anti-PDL1 mAb
11. Systemic application of glucocorticoids or immunosuppressants within 2 weeks prior to the start of the trial. Inhaled corticosteroids and mineralocorticoids are allowed
12. Hormone use contraindications。
13. severe cardiovascular disease, myocardial infection or cerebrovascular accident, arrhythmia, unstable angina within 3 months before the start of the test
14. Uncontrollable increase in blood pressure or elevated blood sugar
15. History of other malignant tumors 5 years ago, except for cervical cancer in situ, non-melanoma skin cancer or stage I uterine cancer
16. Known central nervous system metastasis
17. ≥ NCI CTCAE Level 2 Peripheral Neuropathy
18. serum albumin is less than 2.5 g/dL
19. uncontrollable or symptomatic hypercalcemia
20. Infections requiring antibiotics within 14 days prior to the start of the test
21. chronic enteritis
22. clinically significant active gastrointestinal bleeding
23. Non-diagnostic surgery within 4 weeks prior to the start of the trial 24 There is evidence of the need to limit any other disease using the test drug

25. Participate in other tests within 30 days before the start of the test, or plan to participate in other tests during the test. Accept other experimental drugs within 28 days before the start of the test 26. Women who are pregnant or lactating, or women who are planning to become pregnant within 5 months of the end of treatment. Women of childbearing age are required to undergo a blood pregnancy test within 7 days prior to the start of the trial.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2020-01-20 (Actual); Primary Completion 2024-01-31 (Actual); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
pathological complete response (pCR) rate | up to 2 year
  the rate of no residual tumor cells in both the excised gastric cancer and lymph node (ypT0N0)

SECONDARY OUTCOMES:
Objective Response Rate (ORR) | up to 2 year
  Defined as the proportion of patients with a documented complete response, and partial response (CR
  + PR )
Overall survival(OS) | up to 2 year
  From date of randomization until the date of death from any cause
safety | up to 2 year
  adverse events in patients during the neoadjuvant treatment phase
Disease Free Survival（DFS） | up to 2 year
  The time from the start of randomization to the first tumor recurrence/metastasis or the death of the subject for any reason

CONTACTS AND LOCATIONS:
Overall Officials: Suxia Luo, Principal Investigator — Henan Cancer Hospital
Locations (1):
- Henan Cancer Hospital, Zhengzhou, Henan, China